CLINICAL TRIAL: NCT00963703
Title: Treatment of TNFa Naive Patients With Poor Prognosis Rheumatoid Arthritis Using Rituximab: A Pilot Study Evaluating Synovial Outcomes
Brief Title: Treatment of TNFa Naive Patients With Poor Prognosis Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Dr. Hani El-Gabalawy, Arthritis Centre, Unversity of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2007:160
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab 1000 mg Intravenously day 1 and day 15

SUMMARY:
The purpose of this study is to determine how well Rituximab works in early stages of disease and the effects it has on an inflamed joint and blood cells.

This will allow the investigators to get a better understanding of how this treatment affects the inflamed joints of rheumatoid arthritis (RA) patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented rheumatoid arthritis by ACR criteria
* Disease duration < 5 years
* May have previously been treated with methotrexate,hydroxychloroquine or sulfasalazine, either as a single DMARD or in combination
* Tender joint count >= 6, swollen joint count >= 6, and one must be a knee
* Corticosteroids <= 10 mg per day permitted on stable doses for at least 4 weeks
* Patients must consent to 2 arthroscopic synovial biopsy procedures

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to monoclonal antibodies
* Previous treatment with Rituximab
* Previous treatment with Arava
* Injected with steroids within 4 weeks of day 1 of study
* Treatment with any investigational agent within 4 weeks of day of study
* Any severe or significant medical condition or disease or known active infection
* Pregnancy or nursing at present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To define the synovial effects of rituximab treatment in TNFa naive patients with early rheumatoid arthritis | Biopsies of inflamed joint at beginning and at week 8 of study

SECONDARY OUTCOMES:
To define the effects of rituximab treatment on the phenotype and function of peripheral blood T and B cells | Collected at beginning of study and week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Arthritis Centre, University of Manitoba, Winnipeg, Manitoba, Canada